CLINICAL TRIAL: NCT01211080
Title: Open-label, Uncontrolled Study of the Off Label Use of Propranolol for Infancy Hemangiomas to Identify Side Effects
Brief Title: Off Label Use of Propranolol for Infancy Hemangiomas
Acronym: PIHS
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Carsten Engelmann, Oberarzt, Hannover Medical School
Other Study IDs: AB 3
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Hemangioma
Keywords: infancy hemangioma; propranolol; study design; side effects; safety
MeSH Terms: conditions — Hemangioma | interventions — Propranolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Threatening hemangioma: The group with cosmetically threatening of functionally threatening hemangiomas warranting active treatment according to our usual criteria (location face, hands, feet with a strong growth tendency and below age of 8 months)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Propranolol 2mg/kg/day divided to three oral doses with or without concomitant physical therapy (cryotherapy, laser)

SUMMARY:
Propranolol use for infancy hemangiomas is of world wide interest due to low cost and presumed efficacy. The investigators hypothesized that the drug ist highly active against growing hemangiomas in problematic sites and that there are little side effects.

This observational study was undertaken in an uncontrolled fashion to determine sample size, design and and tools for a later randomized controlled trial on propranolol versus physical therapy (i.e.cryotherapy) which is the most prevalent treatment for the condition. During this initial series side effects and relevant design aspects became evident which warrant expedited reporting.

DETAILED DESCRIPTION:
Treatment modalities: The investigators employed the "best-guess"-dose from the literature at 2 mg/kg/day divided into three daily oral administrations. Individualized capsules were manufactured from Propranolol tablets by the hospital pharmacies and dissolved in sweetened tea before use. Treatment was started at 1mg/kg/day and routinely increased after 24 hrs. or later when three subsequent doses had been tolerated without bradycardia (< 70 bpm when sleeping) or other unwanted events. No other medical treatment was admitted. Physical treatment (cryotherapy, interstitial laser) was administered in parallel to propranolol in 16 patients with threatening hemangiomas (severe impediments to function or cosmesis requiring immediate reduction).

Surveillance and adverse event (AE) reporting:

Pretreatment monitoring included a 24 hr ECG (in KKB a 2 minute rhythm strip), pulse, blood pressure, fasting blood glucose and echocardiography. All patients were kept at a cardiac monitor. Blood pressure was monitored 6 hourly and blood glucose was assayed twice with each new dose at one hour after drug ingestion. If the patient has had 3 full doses the investigators repeated the 24 hr ECG and the echocardiography. Bradycardia and Hypotension events were defined according to the age dependent standards , Side effects/adverse events were defined according to ICH guidelines and screened for as events leading to either a physician contract and a medical measure (dose reduction, ß-mimetic or other medication).

Lesion evaluation:

Hemangioma size was measured with calipers before and after the completed therapy at the end of the 8th month of life. Thickness was checked with a 7.5 mHz linear array pediatric probe.

For evaluation of their cosmesis the lesions were documented with 2 photos each (white balanced flash and ambiance light) before and after treatment (standardized to 30 cm distance, circa 2 Mb resolution). Images were shown at the same week to 3 examiners being unaware whether images were taken pre- or post treatment. This was repeated twice at two weeks interval. As there is no validated hemangioma specific assessment tool a rating form was compiled in an expert discussion from validated scar and burns scales: Categorical items included "Vascularity" and "Height" from the Vancouver Scar Scale , "Irregularity" from the Hamilton burn scar rating form for photographic analysis and the "matte/shiny" classification from the Manchester Scar Scale . A 10 cm plastic surgery visual analogue scale provided non-categorical data on overall appearance.

ELIGIBILITY:
Inclusion Criteria:

Infants with "problematic" true infantile hemangiomas (potentially disfiguring hemangiomas in the face, functional threatening hemangiomas of hands, feet, genitalia)> 4 weeks and < 8 months of age.

Exclusion Criteria:

"Uncomplicated" Hemangiomas (trunk, extremities), infants with heart disease, known arrhythmias, bronchoobstructive disease, known hypoglycaemia events.

Ages: 1 Month to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Tertiary and Secondary Pediatric Surgery Referral unit Secondary Care Pediatrics Unit
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Cosmesis of the lesion and surrounding skin | Completed 8 months of life
  Post treatment cosmetic and defiguration result with a hemangioma specific rating tool for categorical (color, vascularity, height, matte/shiny) and non-categorical data (visual analogue scale for overall appearance) from the Vancouver Burn Scar Scale, the Manchester Scar Scale and the Hamilton Burn scar scale by 3 examiners.
Side effects | Completed 8th month of life
  Number of Participants with Adverse Events in the cardiovascular, bronchopulmonary and metabolic system as a Measure of Safety and Tolerability

SECONDARY OUTCOMES:
hemangioma size | completed 8 th month of life
  Size is measured with calipers and ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Carsten R Engelmann, MD PhD, Principal Investigator — Hannover Medical School; Benno M Ure, Prof., Study Director — Hannover Medical School
Locations (3):
- Germany (3):
  - Pediatric Surgery, Kinderkrankenhaus Bult, Hanover, Hannover
  - Pediatric Surgery, Hannover Medical School, Hanover, Lower Saxony
  - Kinderzentrum Klinikum Hildesheim, Hildesheim, Lower Saxony

REFERENCES:
- [Background] Holland KE, Frieden IJ, Frommelt PC, Mancini AJ, Wyatt D, Drolet BA. Hypoglycemia in children taking propranolol for the treatment of infantile hemangioma. Arch Dermatol. 2010 Jul;146(7):775-8. doi: 10.1001/archdermatol.2010.158. PMID 20644039
- See also: university web site/english — http://www.mh-hannover.de/index.php?id=2&L=1